CLINICAL TRIAL: NCT03401177
Title: The Effect of NSAIDs in the Early Phase of Achilles Tendinopathy
Brief Title: Treatment of Early Phase Achilles Tendinopathy - the Effect of NSAIDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Nikolaj Mølkjær Malmgaard-Clausen, Medical Doctor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BBH-137
Record Dates: First submitted 2017-12-19; First posted 2018-01-17 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Tendon Injuries; Achilles Tendinopathy; Inflammation
MeSH Terms: conditions — Tendon Injuries; Inflammation | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naproxen & Heavy resistance training (Experimental): Naproxen: 500 mg x 2 daily for 7 days, HRT: 3 months physiotherapy guided training.
  Interventions: Drug: Naproxen 500 Mg; Other: Heavy resistance training
- Placebo & Heavy resistance training (Placebo Comparator): Placebo oral tablet: pill manufactured to mimic naproxen tablet x 2 daily for 7 days, HRT: 3 months physiotherapy guided training.
  Interventions: Drug: Placebo Oral Tablet; Other: Heavy resistance training

INTERVENTIONS:
Drug: Naproxen 500 Mg — Naproxen is used as a tool to dampen the inflammation thought to be present in early phase Tendinopathy
  Other Names: Naproxen-E Mylan
  Arms: Naproxen & Heavy resistance training
Drug: Placebo Oral Tablet — Placebo is used, to provide a control to the active group.
  Other Names: Placebo
  Arms: Placebo & Heavy resistance training
Other: Heavy resistance training — Heavy slow resistance training - used in both groups subsequent to the initial week of NSAID or placebo treatment.
  Other Names: HRT

SUMMARY:
this study evaluates the addition of initial short term NSAID treatment to physiotherapy prescribed exercise treatment in patient with early phase tendinopathy. Half of the participants will initially receive NSAID (naproxen) for 7 days, while the other half will receive a placebo, where after both groups will be subjected to 3 months heavy slow resistance training.

DETAILED DESCRIPTION:
NSAID is effective in short term pain relief in musculoskeletal disorders, but little is known about the long-term effect in early phase tendinopathy, when used as a supplement to treatment as usual, namely heavy slow resistance training and training load reduction. In this study, NSAIDs will be used, which works through COX inhibition, which again inhibits Prostaglandins, in this way investigators attempt to dampen the initial inflammation and pronounced cell activity that is thought to be present in early phase tendinopathy. With this project, it will be attempted to investigate whether initial dampening adds to the effect achieved through heavy load resistance training, which is thought to stimulate structural repair and regeneration in the tendon, by applying appropriate load to the tendon tissue, thereby stimulating the tendon cells to repair and regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Activity related pain in the achilles tendon
* Palpation pain in the achilles tendon
* Onset of symptoms within the last 3 months

Exclusion Criteria:

* Previous injury in the achilles tendon on the ipsilateral side.
* Recent infection around the achilles tendon
* Previous surgery in the achilles tendon.
* Contraindications for NSAID treatment.
* NSAID treatment for the current injury
* Medication with NSAID interaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles (VISA-A) | 0-3 months
  Standardised score of functional capability, in patient with achilles tendinopathy. Total score will be reported; scale (0-100). 100=full functional capacity 0=poor functional capacity.

SECONDARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles (VISA-A) | 0-1 week; 0-12 months
  Standardised score of functional capability, in patient with achilles tendinopathy.
  Total score will be reported; scale (0-100). 100=full functional capacity 0=poor functional capacity.
Weight | 0-3 months
  Weight (kg)
Height | 0-3 months
  Height (cm)
Magnetic Resonance Imaging (MRI) - scannings | 0-3 months
  3 Tesla MRI scanning of the achilles tendon.
Ultrasonography -Power doppler | 0-1 week; 0-3 months
  For measuring tendon vascularisation, area with power doppler signal (cm^2)
Ultrasonography - Greyscale | 0-1 week; 0-3 months
  Greyscale ultrasound for measuring tendon thickness (mm)
Questionnaires - activity (time consumption) | 0-1 week; 0-3 months; 0-12 months
  Questions on physical activity: time consumption (hours/week)
  Hours of training/week;
  Hours of training applying load on the achilles tendon/week; Scale (continues)
Questionnaires - activity (number of sessions) | 0-1 week; 0-3 months; 0-12 months
  Questions on physical activity: number of sessions/week
  Number of training sessions/week.
  Number of training sessions applying load on the achilles tendon/week; Scale (continues)
Questionnaires - activity (intensity) | 0-1 week; 0-3 months; 0-12 months
  Questions on physical activity intensity:
  time consumption for strenuous activity (hours/week).
Questionnaires - Numerical Rating Scale (NRS) - Pain | 0-1 week; 0-3 months; 0-12 months
  Questions on pain, both during activity and during rest.
  Pain during activity, (NRS); Scale (0-10)
  Pain after activity, (NRS); Scale (0-10)
  Pain at rest, (NRS); Scale (0-10)
  Pain I the morning, (NRS); Scale (0-10)
  Maximal pain during the past week, (NRS); Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjær, Professor, Study Director — Institute of Sports Medicine, Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malmgaard-Clausen NM, Jorgensen OH, Hoffner R, Andersen PEB, Svensson RB, Hansen P, Nybing JD, Magnusson SP, Kjaer M. No Additive Clinical or Physiological Effects of Short-term Anti-inflammatory Treatment to Physical Rehabilitation in the Early Phase of Human Achilles Tendinopathy: A Randomized Controlled Trial. Am J Sports Med. 2021 Jun;49(7):1711-1720. doi: 10.1177/0363546521991903. Epub 2021 Mar 15. PMID 33719579